CLINICAL TRIAL: NCT00617149
Title: Effect of Regular Exercise in Prevention of Excessive Weight Gain in Pregnancy. A Single Blind Randomized Controlled Trial
Brief Title: Effect of Regular Exercise in Prevention of Excessive Weight Gain in Pregnancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Responsible Party: Lene AH Haakstad, Msci, Ph.D student, Exercise scientist, Norwegian School of Sport Sciences, Department of Sport Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-05208 (REK); 17804/2/KH (NSD)
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Pregnancy; Excessive Weight Gain
Keywords: exercise,; excessive weight gain during pregnancy
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Supervised exercise for the prevention high weight gain — Each session starts with ca 5 minutes warm up, followed by 30 minutes of aerobic activity, including cool down. This is followed by 15 minutes of strength training of the upper and lower limbs, and special focus on the deep abdominal stabilization muscles. The last 5 minutes contains stretching, relaxation and body awareness exercises. The exercise-program follows the ACOG exercise prescription, and all aerobic activities will be performed at moderate intensity (60-70% of maximal heart rate), measured by ratings of perceived exertion at 11-14 (somewhat hard) on the 6-20 Borg's rating scale. Control-participants are neither encouraged nor discouraged from exercising.
  Other Names: exercise, excessive weight gain, pregnant women

SUMMARY:
Background:

Use of variable definitions of exercise and disparate results, emphasize the need of proper randomized controlled trials examining the relationship between physical activity and weight development during pregnancy. So far, only few intervention studies aiming at weight management during pregnancy have been performed (Gray-Donald et al., 2000,Olson et al., 2004,Polley et al., 2002,Kinnunen et al., 2007). Moreover, most of these interventions have focused on how gestational weight gain may be altered through individual counselling combining diet and exercise habits, rather than supervised training. Search on PubMed revealed no randomized controlled trial where the main outcome was to investigate how the effect of supervised structured exercise may reduce the proportion of women gaining more weight than optimal. The aim of the present study is to assess whether a 12-week aerobic exercise program during pregnancy can prevent excessive gestational weight gain.

Method:

This is a single blind randomized controlled trial to evaluate the effects of a structured, supervised aerobic exercise program on weight gain stabilization in primiparous pregnant women. The aim is to include 100 women. Interested women eligible for the present study will be invited to a pre-test including interview and assessments at the university. The women are examined three times during the study period. The first visit is between 12 and 24 weeks of gestation, the second at week 36-38 and the last 8-12 week after delivery. The exercise program consists of supervised exercise for 60 minutes, performed at least 2 times per week, for 12-16 weeks. Compliance with the training protocol is controlled by the instructors and registrations in the womens personal training diary

DETAILED DESCRIPTION:
Background:

Data from population-based surveys and longitudinal observational studies generally support that inactive men and women have higher body weight and BMI than physically active adults (US Departmentof Health and Human Services, 1996,Williamson et al., 1993,Sherwood et al., 2000,Anderssen et al., 2007). Studies examining the impact of exercise on maternal weight gain are varied and limited. Two different meta- analysis's found no difference in maternal weight gain between exercisers and non-exercisers (Kramer, 2002,Lokey et al., 1991). In a review from 2004 it is suggested that women who exercise before pregnancy and continue to do so during pregnancy tend to weigh less and gain less weight that controls (Siega-Riz et al., 2004). A recent study of Haakstad et al (Haakstad et al., 2007) found that women who continued to exercise regularly in the 3rd trimester had significantly lower total weight gain. In addition, women reporting high exercise frequency in the 3rd trimester ( ≥ 4 times per week), the proportion exceeding IOM's weight gain recommendations was significantly lower compared to women exercising less frequently (1-3 times per week)(Haakstad et al., 2007). These results indicate that there may be a dose-respons relationship, with higher levels of exercising being more effective than moderate and low levels for the prevention of high maternal weight gain.

So far, only few intervention studies aiming at weight management during pregnancy have been performed (Gray-Donald et al., 2000,Olson et al., 2004,Polley et al., 2002,Kinnunen et al., 2007). Moreover, most of these interventions have focused on how gestational weight gain may be altered through individual counselling combining diet and exercise habits, rather than supervised training. Search on PubMed revealed no randomized controlled trial where the main outcome was to investigate how the effect of supervised structured exercise may reduce the proportion of women gaining more weight than optimal. The aim of the present study is to assess whether a 12-week aerobic exercise program during pregnancy can prevent excessive gestational weight gain.

Method:

Participants This is a single blind randomized controlled trial to evaluate the effects of a structured, supervised aerobic exercise program on weight gain stabilization in primiparous pregnant women. Participants will be recruited via health practitioners (physicians, midwifes), articles and advertisement in the newspapers, official websites for pregnant women, through flyers and word of mouth. The aim is to include 100 women. With power = 0.85 and alfa = 5%, the present study is designed to detect a standardized difference in total weight gain of 0.6. Assuming that the standard deviation of weight gain is 5 kilos, then the actual weight gain has to be ∆= 3 kilos.

Inclusion/exclusion At first contact by phone, the aim and implications of the study are explained and the eligibility criteria are checked. Primiparous women who have not participated in a structured exercise program, including significant amounts of walking for the past six months is eligible for the trial. Other inclusion criteria are ability to read, write and speak Norwegian, and to be within their first 24 weeks of pregnancy. Exclusion criteria is severe heart disease, pregnancy induced hypertension, history of more than two miscarriages, persistent bleeding after week 12 of gestation, poorly controlled thyroid disease, poorly controlled pre-eclampsia and other diseases that could interfere with participation (Artal and O'Toole, 2003). In addition, all women who live to far from the university to be able to attend weekly training groups will be ineligible.

Procedure and outcome measures Interested women eligible for the present study will be invited to a pre-test including interview and assessments at the university. All visits are accomplished during daytime and at normal working hours. The women are examined three times during the study period. The first visit is between 12 and 24 weeks of gestation, the second at week 36-38 and the last 8-12 week after delivery. Each visit lasts about 60-75 minutes. There is no induction to the exercise program before gestation week 12.

At the first appointment, the principal investigator (LH) completes an initial interview and health screening with all participants. The requirements of the study are explained and possible contraindications for exercise are identified again. Data from the Pregnancy Health Card is registered. The baseline questionnaire covers demographic information (e.g. age, pregnancy week, smoking habits, education, occupation), assessment of daily life physical activity and sedentary behaviour (at work, in transportation and household). In addition, there is registration of pregnancy complications (e.g. pelvic girdle and low back pain, urinary incontinence, high blood pressure, pre-eclampsia, vomiting, fatigue). The second questionnaire is self administrated and includes questions about perceived quality of life and health status the last four weeks. Finally, the women's pre-pregnancy weight is registered and hight and weight is measured using a digital beam scale. Anthropometric estimation of maternal body composition is assessed by Holtain caliper, measuring left side skinfold thickness of the triceps, abdomen and thigh. Each measurement is done twice and held for 5-10 seconds. A mean value of the two is computed. If the two skinfold assessments differ more than 2mm, the skinfold is measured a third time and the mean of the three values are calculated.

The same assessments described above are obtained at the second visit (week 36-38 of gestation). At the third and last visit (8-12 week postpartum), the women will also report infant birth weight and complications during delivery. The women are asked to bring health the journal from the hospital and the Infant Health Card

All subjects will complete two sub maximal step treadmill tests. One test immediately after randomization and the second test at week 36-38 of gestation. The main sub maximal functional outcome is oxygen uptake and lactate measurements. After adjustments to the treadmill, nose clip and mouthpiece, all participants start walking on an initial speed of 4.5 km/h. The inclination will elevate each fourth minutes with exactly 4%. Blood pressure, heart rate and rating of perceived exertion (6-20 scale) (Borg, 1970) are measured during the last two minutes of every step after steady state is reached based on stable oxygen uptake measurements. Capillary blood sample for measuring blood lactate is assessed in the 30 second pause after each step. The test is determined after 12-20 minutes when the subjects blood lactate concentration rise about 1.5 mMol∙L-1 above resting level or perceive physical exertion between 15-17 (Borg scale) and/or a heart rate < 85% of expected maximal heart rate. The same exercise physiologist will perform both tests.

All participants gave written consent to participate, and the procedures to be followed are in accordance with the ethical standards of the responsible regional committee on human experimentation and adhered to the World Medical Association Declaration of Helsinki. The project was received and approved by The Committee for Medical Research Ethics, Southern Norway, Oslo, Norway, on 20 February 2006 (reference number S-05208). Additionally, the Norwegian Social Sciences Data Services (NNT) provided licence to store and register individual health information (reference number 17804/2/KH). All data will be stored and locked in a fireproof cabinet and are in accordance with requisitions from NNT. The inclusion of women to the trial started in Sept 2007 and will continue till 100 participants are randomly allocated to the exercise and control groups. All follow-up procedures are expected to finish within Mars 2009. There is no financial compensation to the participants.

Randomization procedure The randomization procedure will take place after determination of eligibility, completed baseline examination and measurement of primary outcome variables. Based on a statistical randomization computer program, an independent person is assigning the participants to the two groups. The participants will be informed not to reveal any information about which group they are assigned for to the principal investigator (LH). The principal investigator is not involved in the training of the women and is blinded to group allocation while making the outcome measures and plotting all data. It has not been considered ethically incorrect to use a control group not receiving treatment in present study.

Exercise program The exercise program consists of supervised exercise for 60 minutes, performed at least 2 times per week, for 12-16 weeks. Since most participants are working full time, the exercise groups are arranged in the evening. Each session starts with ca 5 minutes warm up, followed by 30 minutes of aerobic activity, including cool down. This is followed by 15 minutes of strength training of the upper and lower limbs, and special focus on the deep abdominal stabilization muscles (the transversus abdominus muscle, pelvic floor and back muscles). The last 5 minutes contains stretching, relaxation and body awareness exercises. Aerobic exercises include only low impact exercise (no jumping or running). Step length and body rotations are reduced to a minimum, and crossings of legs and sharp and sudden changes of position are avoided. The exercise-program follows the ACOG exercise prescription, and all aerobic activities will be performed at moderate intensity (60-70% of maximal heart rate), measured by ratings of perceived exertion at 11-14 (somewhat hard) on the 6-20 Borg's rating scale. The exercise program is choreographed and led by certified aerobic instructors, and each session includes maximum 25 participants. In addition to joining the scheduled aerobic classes, all women are motivated to include 30 minutes of moderate self-imposed physical activity on the rest of the week-days. They will also be advised to incorporate short bouts of activity into their daily schedules. For example, participants are encouraged to walk instead of drive short distances and to use stairs instead of elevators. The participants are asked to keep daily records of their minutes of physical activity. Compliance with the training protocol is controlled by the instructors and registrations in the womens personal training diary. Control-participants are neither encouraged nor discouraged from exercising.

Statistical analysis Analysis will be completed to assess the effects of the intervention on two primary and five secondary outcomes: Primary outcomes are overall weight gain during pregnancy and proportion of participants exceeding weight gain above IOM recommendations. Secondary outcomes are pregnancy complications, relationship between oxygen consumption, heart rate and blood lactate concentration at submaximal work loads, infant birth weight, length of labour and complications during delivery.

The principal analysis will be done on an intention to treat basis. Missing values are carried forward by their baseline values. The primary dependant variables are total weight gain and the proportion of women who exceed the IOM recommendations. Average total weight gain is compared between the two groups and the possible difference is tested using two-sided independent sample t-test. The group differences in the proportion of participants who gained weight above the IOM guidelines are tested by using two-sided X2-test.

The secondary outcomes; self-report of complications during pregnancy and delivery, as well as number of high birth weight infants (≥4200 g) (Skjaerven et al., 2000,Orskou et al., 2003) will be compared between the intervention and control group and tested using X2-test or Fisher's exact test. The two-sided independent sample t-test is used to test the difference in submaximal cardiorespiratory capacity, gestation weeks at delivery, infant's birth weight and duration of labour. In all statistical analysis, level of statistical significance is set at p<0.05. Professor of biostatistics, Ingar Holme, Norwegian Scholl of Sport Science, is advising the present study.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women who have not participated in a structured exercise program, including significant amounts of walking for the past six months are eligible for the trial.
* Other inclusion criteria are ability to read, write and speak Norwegian, and to be within their first 24 weeks of pregnancy.

Exclusion Criteria:

* Severe heart disease
* Pregnancy induced hypertension
* History of more than two miscarriages
* Persistent bleeding after week 12 of gestation
* Poorly controlled thyroid disease
* Poorly controlled pre-eclampsia and/or other diseases that could interfere with participation (Artal and O'Toole, 2003)
* In addition, all women who live to far from the university to be able to attend weekly training groups will be ineligible

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Primary outcomes are overall weight gain during pregnancy and proportion of participants exceeding weight gain above IOM recommendations. | week 36-38 of pregnancy

SECONDARY OUTCOMES:
Secondary outcomes are pregnancy complications, relationship between oxygen consumption, heart rate and blood lactate concentration at submaximal work loads, infant birth weight, length of labour and complications during delivery. | week 36-38 of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Lene Haakstad, PhD student, Principal Investigator — Norwegian School of Sport Science
Locations (1):
- Norwegian School of Sport Science, Oslo, Norway

REFERENCES:
- [Derived] Haakstad LAH, Bo K. The marathon of labour-Does regular exercise training influence course of labour and mode of delivery?: Secondary analysis from a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2020 Aug;251:8-13. doi: 10.1016/j.ejogrb.2020.05.014. Epub 2020 May 12. PMID 32460116
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] Halvorsen S, Haakstad LA, Edvardsen E, Bo K. Effect of aerobic dance on cardiorespiratory fitness in pregnant women: a randomised controlled trial. Physiotherapy. 2013 Mar;99(1):42-8. doi: 10.1016/j.physio.2011.11.002. Epub 2012 Apr 3. PMID 23186730
- [Derived] Haakstad LA, Bo K. Exercise in pregnant women and birth weight: a randomized controlled trial. BMC Pregnancy Childbirth. 2011 Sep 30;11:66. doi: 10.1186/1471-2393-11-66. PMID 21961534
- [Derived] Bo K, Haakstad LA. Is pelvic floor muscle training effective when taught in a general fitness class in pregnancy? A randomised controlled trial. Physiotherapy. 2011 Sep;97(3):190-5. doi: 10.1016/j.physio.2010.08.014. Epub 2011 Feb 4. PMID 21820536